CLINICAL TRIAL: NCT04484740
Title: Penetration of the Innovative Antibiotic Gepotidacin Into Prostate and Tonsillar Tissue.
Acronym: AB-Direct
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C19-28; 2019-004308-37 (EudraCT Number)
Record Dates: First submitted 2020-07-10; First posted 2020-07-24 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Gonorrhea; Infection, Bacterial
Keywords: tissue pharmacokinetics; gepotidacin; microdialysis
MeSH Terms: conditions — Gonorrhea; Bacterial Infections | interventions — gepotidacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gepotidacin (Experimental)
  Interventions: Drug: Gepotidacin

INTERVENTIONS:
Drug: Gepotidacin — Single oral dose of 1500 mg gepotidacin

SUMMARY:
Gepotidacin is a new antibiotic that may potentially be used to treat prostatic infections and pharyngeal gonorrhoea. To date, no data exists on gepotidacin pharmacokinetics in those tissues. The present study is being carried out to determine concentrations of gepotidacin in plasma, prostate and tonsillar tissue of patients undergoing radical prostatectomy (RPE) for localized prostate, simple prostatectomy (PE) for benign prostate hyperplasia (BPH) or tonsillectomy (TE). This will contribute to a more complete understanding of the drug's penetration to its site of action.

DETAILED DESCRIPTION:
A single dose of 1500 mg gepotidacin will be administered to patients who will undergo radical prostatectomy (RPE) or simple prostatectomy (PE) and patients undergoing tonsillectomy (TE). The individual time-points of gepotidacin administration will be chosen to ensure that the time-point of tissue removal corresponds with one of six different sampling time-points, as closely as possible.

After study drug administration RPE or TE will be performed according to clinical routine.

Subsequently, microdialysis (MD) probes will be inserted in the removed tissue (tonsillar or prostate tissue) ex-vivo and MD will be performed to determine unbound drug concentrations in the tissue.

Plasma PK samples will be collected just before study drug administration and up to 48h after administration of gepotidacin.

Since MD provides the concentration of the unbound fraction of gepotidacin, for comparison we will calculate the unbound fraction of the concentration values obtained through blood sampling. To this end, we will determine the protein binding using ultrafiltration for each subject at the time-point closest to the Cmax. The individual protein binding can then be used to calculate the unbound plasma fraction of gepotidacin. This will allow to transform the plasma PK data to the same scale as the microdialysis data.

Samples will be analysed using non-compartmental analysis (NCA) for plasma concentrations and population pharmacokinetic models (PopPK) for tissue concentrations pooled with plasma concentrations.

ELIGIBILITY:
Inclusion Criteria:

Cohort A only:

* Clinically localized prostate cancer or benign prostate hyperplasia
* Male patient scheduled for prostatectomy

Cohort B only:

* Male or female patient scheduled for complete tonsillectomy
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP) or
  * Is a WOCBP with a highly sensitive negative pregnancy test

Both Cohorts:

* Age: above 18 years
* Body weight ≥40 kg and body mass index (BMI) within the range 18.5 - 32.0 kg/m2
* A signed and dated written informed consent form
* The subject is able to understand and willing to comply with protocol requirements and timetables, instructions and protocol-stated restrictions
* Negative serology (human immunodeficiency virus, hepatitis B-AG and C-AB) at screening
* Patient with a social security or health insurance (if applicable according to the local regulation)

Exclusion Criteria:

Cohort A only:

• Any concerns of the investigator or the treating urologists that the participation in the study might impair histological assessment of the prostate tissue such as (but not limited to): lack of representative histology via previous biopsy AND inability to safely insert microdialysis probes in tissue with sufficient distance to the tumor (e.g. large or diffuse tumor, lack of MRI or PET image to locate tumor within the organ).

Cohort B only:

* Pregnancy
* Women of childbearing potential who are not employing adequate contraceptive measures
* Accepted contraceptive measures are (have to be employed for at least 30 days prior to dosing until one week after the final examination):

  * intrauterine device
  * intrauterine hormone-releasing system
  * implantable progestogen-only hormone contraception associated with inhibition of ovulation
  * combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal, injectable)
  * progestogen-only hormone contraception associated with inhibition of ovulation (oral, injectable)
  * condoms
  * sexual abstinence
  * surgical sterilization
* Acute tonsillitis or peritonsillar abscess
* History of peritonsillar abscess
* Tonsillectomy for cervical lymph node metastasis of cancer of unknown primary

Both Cohorts:

• Individuals deprived of liberty and protected persons (under guardianship or curatorship).

Medical Conditions

* Clinically significant abnormality in the past medical history or at the Screening physical examination that in the investigator's opinion may place the participant at risk or interfere with outcome variables of the study. This includes, but is not limited to, history or current cardiac, hepatic, renal, neurologic, gastrointestinal (GI), respiratory, hematologic, or immunologic disease.
* Any surgical or medical condition that may be aggravated by inhibition of acetylcholinesterase, such as:

  * Poorly controlled asthma or chronic obstructive pulmonary disease at baseline and, in the opinion of the investigator, not stable on current therapy
  * Acute severe pain, uncontrolled with conventional medical management
  * Active peptic ulcer disease
  * Parkinson disease
  * Myasthenia gravis
  * A history of seizure disorder requiring medications for control (this does not include a history of childhood febrile seizures)
* Any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study intervention, or any other condition that may place the participant at risk, in the opinion of the investigator.
* Within 2 months before Screening, either a confirmed history of Clostridium difficile diarrhoea infection or a past positive C. difficile toxin test.
* Uncompensated heart failure
* Severe left ventricular hypertrophy
* History of significant vasovagal and/or syncopal episodes or episodes of symptomatic bradycardia
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of drug and/or alcohol abuse within 6 months before screening, as determined by the investigator
* History of sensitivity to any of the study drug, components thereof, or a history of drug or other allergy that, in the opinion of the investigator contraindicates their participation.
* Subject is taking QT-prolonging drugs or drugs known to increase the risk of torsades de points (TdP) per the www.crediblemeds.org "Known Risk of TdP" category at the time of screening that cannot be discontinued. If discontinued they should be discontinued at screening and can be resumed after the last PK sample.
* Subject is taking strong cytochrome P450 enzyme 3A4 (CYP3A4) inhibitors CYP3A4 that cannot be discontinued. If discontinued, they should be discontinued at a minimum of 12 hours or 5 half-lifes from the scheduled gepotidacin dose and can be resumed after the last PK sample.
* Subject is taking strong P glycoprotein (P-gp) inhibitors that cannot be discontinued. If discontinued, they should be discontinued at a minimum of 12 hours or 5 half-lifes from the scheduled gepotidacin dose and can be resumed after the last PK sample.

Prior/Concurrent Clinical Study Experience

• Previous exposure to gepotidacin. Participant has participated in a clinical trial and has received an investigational product prior to gepotidacin administration within 30 days, 5 half-lives, or twice the duration of the biological effect of investigational product (whichever is longer) Non-interventional studies are excepted.

Diagnostic assessments

* Alanine aminotransferase (ALT) >1.5 × upper limit of normal (ULN).
* Bilirubin >1.5 × ULN (isolated bilirubin >1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* History of any kidney disease or current or chronic history of impaired renal function as indicated by an estimated creatinine clearance <60 mL/min.
* History of regular alcohol consumption within 6 months of screening defined as an average weekly intake of >21 units (or an average daily intake of >3 units) for males or an average weekly intake of >14 units (or an average daily intake >2 units) for females. One unit is equivalent to 270 mL of full strength beer, 470 mL of light beer, 30 mL of spirits, or 100 mL of wine.
* History of regular use of more than 10 cigarettes or equivalent per day.
* Clinically significant abnormal findings in serum chemistry, hematology, or urinalysis results obtained at screening at investigators discretion
* Baseline corrected QT interval using the Fridericia formula (QTcF) of >450 msec.

Other Exclusions

* Participant has donated blood in excess of 500 mL within 12 weeks prior to dosing or participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* Participant is unable to comply with all study procedures, in the opinion of the investigator.
* Participant should not participate in the study, in the opinion of the investigator or sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-05-27 (Actual); Study Completion 2023-05-27 (Actual)

PRIMARY OUTCOMES:
area under the concentration time curve (AUC) from zero to last observed concentration (AUC0-t) in tissue | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in tissue calculated using a population pharmacokinetic model
AUC from zero to infinity (AUC0-∞) in tissue | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in tissue calculated using a population pharmacokinetic model
maximum drug concentration (Cmax) in tissue | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in tissue calculated using a population pharmacokinetic model
half-life (t1/2) in tissue | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in tissue calculated using a population pharmacokinetic model
time to reach maximum drug concentration (tmax) in tissue | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in tissue calculated using a population pharmacokinetic model

SECONDARY OUTCOMES:
area under the concentration time curve (AUC) from zero to last observed concentration (AUC0-t) in plasma | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in plasma calculated using a population pharmacokinetic model
AUC from zero to infinity (AUC0-∞) in plasma | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in plasma calculated using a population pharmacokinetic model
Cmax in plasma | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in plasma calculated using a population pharmacokinetic model
t1/2 in plasma | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in plasma calculated using a population pharmacokinetic model
tmax in plasma | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in plasma calculated using a population pharmacokinetic model
apparent volume of distribution (Vd) in plasma | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in plasma calculated using a population pharmacokinetic model
Clearance (Cl) in plasma | Baseline to 48 hours after drug administration
  Pharmacokinetic parameters in plasma calculated using a population pharmacokinetic model
T>MIC in tissue and plasma (if applicable) | Baseline to 48 hours after drug administration
  PK/PD parameter
Cmax/MIC in tissue and plasma | Baseline to 48 hours after drug administration
  PK/PD parameter
AUC/MIC in tissue and plasma (if applicable) | Baseline to 48 hours after drug administration
  PK/PD parameter
collection of adverse events during study participation | at the final examination (2 to 5 days after study drug administration)
  Drug safety

CONTACTS AND LOCATIONS:
Locations (4):
- MUVienna, Vienna, Austria
- France (3):
  - CHU POITIERS Département ORL, Poitiers
  - CHU POITIERS Département Urologie, Poitiers
  - CHRU TOURS Département Urologie, Tours